CLINICAL TRIAL: NCT01839448
Title: Frequency of Abnormal Glucose Metabolism (Diabetes, Impaired Glucose Tolerance, Impaired Fasting Glucose) in the Immediate Postpartum Period Following Gestational Diabetes Diagnosed Before or After 24 Weeks of Gestation
Brief Title: Abnormal Post-partum Glucose Metabolism After Gestational Diabetes Diagnosed Before or After 24 Weeks of Gestation
Acronym: DG Post-Partum
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2012/VC-01; 2013-A00277-38 (Other: ANSM)
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2018-01

CONDITIONS: Gestational Diabetes; Type 2 Diabetes; Glucose Intolerance
Keywords: post partum diabetes; impaired fasting glucose
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GD diagnosis before 24 weeks: Patients in this group are diagnosed with gestational diabetes (GD) before 24 weeks of amenorrhea by means of a fasting blood glucose test >= 0.92 g/l.
  Intervention: Post-partum oral glucose tolerance test
  Interventions: Biological: Post-partum oral glucose tolerance test
- GD diagnosed at 24 to 28 weeks: Patients in this group are diagnosed with gestational diabetes between 24 and 28 weeks of amenorrhea based on a normal fasting blood glucose level before 24 weeks of amenorrhea AND an abnormal oral glucose tolerance test between 24 and 28 weeks of amenorrhea.
  Intervention: Post-partum oral glucose tolerance test
  Interventions: Biological: Post-partum oral glucose tolerance test

INTERVENTIONS:
Biological: Post-partum oral glucose tolerance test — All patients will have an oral glucose tolerance test at 4 to 12 weeks after the end of pregnancy. Study representatives will contact patients by phone to remind them of the necessity of this test, and its importance for their health.

SUMMARY:
The main objective of the study is to estimate and compare the percentage of patients with abnormal glucose metabolism at 4-12 weeks postpartum between two groups: patients diagnosed with gestational diabetes before or after 24 weeks of pregnancy. Abnormal glucose metabolism is defined as type 2 diabetes, glucose intolerance or impaired fasting glucose.

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare between the two groups:

A. the rate of type 2 diabetes only, glucose intolerance only, impaired fasting glucose only, and patients requiring insulin at 4-12 weeks postpartum

B. rates of maternal and obstetric complications

C. risk factors (age, body mass index, personal history of gestational diabetes or macrosomia, first degree family history of diabetes).

D. For fasting glucose done before 24SA, we will calculate the optimal threshold for predicting abnormal glucose metabolism in the immediate postpartum period among women with gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 10 months of follow-up
* The patient is pregnant and consulting before 24 weeks of amenorrhea AND has at least one of the following risk factors: age > 35 years; body mass index > 25; family history of type 2 diabetes; history of gestational diabetes; history of macrosomia.
* The patient has a fasting blood glucose level >= 0.92 g/l before 24 weeks of amenorrhea OR a fasting blood glucose level < 0.92 g/l before 24 weeks of amenorrhea AND an abnormal oral glucose tolerance test (75 g of glucose) between 24 and 28 weeks of amenorrhea (normal values are set at T0 < 0.92 g/l; T60 < 1.80 g/l; T120 < 1.53 g/l).

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study, with the exception of the following studies: Papillo PMA (RCB 2013-A00538-37), LXRs (RCB 2009-A00968-49), GrossPath (RCB 2014-A01120-47), BAKRI (RCB 2013-A00914-41), OASIS II (RCB 2013-A00773-42), ElastoMAP (RCB 2013-A01148-37), ElastoDéclench (RCB 2014-A00828-39) and UpSideDown (RCB 2014-A01921-46).
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient cannot read French
* The patient has a known history of type 2 diabetes
* The patient is diagnosed with type 2 diabetes during pregnancy (fasting blood glucose level > 1.26 g/l)
* The patient has a contra-indication for a treatment necessary for this study
* The patient is taking chronic or intermittent oral or inhaled corticosteroids, or a β2 agonist treatment for a previous disease or a disease discovered during pregnancy within one week preceding the fasting glucose or oral glucose tolerance test.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of pregnant women consulting before 24 weeks of amenorrhea and who have at least one of the following risk factors: age > 35 years; body mass index > 25; a family history of type 2 diabetes; a history of gestational diabetes or macrosomia.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-03-27 (Actual); Primary Completion 2016-10-12 (Actual); Study Completion 2016-10-12 (Actual)

PRIMARY OUTCOMES:
Presence/absence of abnormal glucose metabolism | 4 to12 weeks post-partum
  Includes type 2 diabetes, glucose intolerance and impaired fasting glucose

SECONDARY OUTCOMES:
Presence/absence of type 2 diabetes | 4 to 12 weeks post partum
Presence/absence of glucose intolerance | 4 to 12 weeks post-partum
Presence/absence of impaired fasting glucose | 4 to12 weeks post-partum
  American definition: defined as between 1 and 1.26 g/l
Presence/absence of impaired fasting glucose | 4 to12 weeks post-partum
  European definition: defined as between 1.1 and 1.26 g/l
Patient requiring insulin: yes/no | 4 to12 weeks post-partum
Presence/absence of complications | 4 to12 weeks post-partum
  This includes a yes/no response for each of the following: caesarean section, hypertension, preeclampsia, urinary tract infection, macrosomia, dystocia, neonatal transfer, respiratory distress, threat of premature birth.
Baby's weight at birth (kg) | 4 to 12 weeks post-partum
Weeks of amenorrhea (duration of pregnancy in weeks/ gestational age) | 4 to 12 weeks post-partum
Patient was older than 35 years of age at beginning of pregnancy? yes/no | baseline (day 0)
Body mass index > 25 at beginning of pregnancy? yes/no | baseline (day 0)
First degree family history of type 2 diabetes? yes/no | baseline (day 0)
History of gestational diabetes? yes/no | baseline (day 0)
History of macrosomia? yes/no | baseline (day 0)
Fasting glucose (g/l) | before 24 weeks of amenorrhea
Oral glucose tolerance test results if necessary | 24 to 28 weeks of amenorrhea

OTHER OUTCOMES:
Age | baseline (day 0)
Body mass index | baseline (day 0)
Number of pregnancies | baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Valéria Cosma, MD, Study Director — Centre Hospitalier Universitaire de Nîmes; Anne-Marie Guedj, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - CH d'Arles - Hôpital Joseph Imbert, Arles
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes

REFERENCES:
- [Result] Cosma V, Imbernon J, Zagdoun L, Boulot P, Renard E, Brunet C, Mares P, Rodier M, Kabani S, Demattei C, Guedj AM. A prospective cohort study of postpartum glucose metabolic disorders in early versus standard diagnosed gestational diabetes mellitus. Sci Rep. 2021 May 17;11(1):10430. doi: 10.1038/s41598-021-89679-2. PMID 34001938